CLINICAL TRIAL: NCT06332300
Title: An Exploratory Clinical Study of Adebelimumab in Combination With Famitinib and Lateral Ventricular Chemotherapy in Patients With Non-squamous NSCLC With Soft Meningeal Metastases Who Have Failed EGFR-TKI Therapy
Brief Title: An Exploratory Clinical Study of Adebelimumab in Combination With Famitinib and Chemotherapy in Patients With NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study drug, Famitinib, was not marketed and the drug was not available.
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADBL-LC-003
Record Dates: First submitted 2024-03-12; First posted 2024-03-27 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebelimumab+famitinib+chemotherapy (Experimental): Adebelimumab in combination with famitinib and lateral ventricular chemotherapy in patients with non-squamous NSCLC with soft meningeal metastases who have failed EGFR-TKI therapy
  Interventions: Drug: Adebelimumab+Famitinib + FOLFIRI+Ariely

INTERVENTIONS:
Drug: Adebelimumab+Famitinib + FOLFIRI+Ariely — Adebelimumab in combination with famitinib and lateral ventricular chemotherapy in patients with non-squamous NSCLC with soft meningeal metastases who have failed EGFR-TKI therapy

SUMMARY:
This study was a single-arm design to explore the efficacy and safety of Adebelimumab in combination with famitinib and lateral ventricular chemotherapy in patients with floppy meningeal metastases from non-squamous NSCLC who have failed EGFR-TKI therapy, and included patients with pathologically confirmed non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
Despite the rapid progress of immune-combination therapy in lung cancer, immune-combination anti-vascular regimens after EGFR-TKI failure have not been explored in NSCLC LM, and further exploration of superior regimens targeting brain metastases is needed. Therefore, we plan to conduct an exploratory clinical study of adebenosumab in combination with famitinib and lateral ventricular chemotherapy in patients with non-squamous NSCLC with soft meningeal metastases who have failed EGFR-TKI therapy, with the aim of providing a more feasible and effective comprehensive treatment strategy for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form (ICF)
2. Aged 18-75 years old, male or female.
3. Histologically or cytologically confirmed EGFR mutation-positive non-squamous NSCLC (International Association for the Study of Lung Cancer (IASLC) 8th edition TNM staging criteria)
4. LM diagnosis confirmed by positive CSF cytology
5. Re-biopsy (histology or cytology or hematology) after treatment failure with at least one EGFR tyrosine kinase inhibitor (EGFR-TKI) suggesting no EGFR-sensitive mutation and possibly other treatments
6. All patients are required to have NSCLC associated with at least 1 LM site identified by the investigator that can be evaluated by MRI scanning and is amenable to repeat evaluation.
7. not required to have received systemic corticosteroids (>10mg/day prednisone or equivalent) within 2 weeks prior to enrollment
8. Expected survival ≥ 12 weeks
9. Vital organ function within 1 week before enrollment meets the following criteria: (1) blood routine: white blood cell (WBC) ≥3.0×109/L; absolute neutrophil count (ANC) ≥1.5×109/L; platelet (PLT) ≥100×109/L; hemoglobin (HGB) ≥9.0 g/Dl (2) Liver function: aspartate transferase (AST) ≤2.5×ULN, alanine aminotransferase (ALT) ≤2.5×ULN. (3) Renal function: serum creatinine ≤1.5×ULN or creatinine clearance rate (creatinine) ≤1.5×ULN; serum bilirubin (TBIL) ≤2.5×ULN, alanine aminotransferase (ALT) ≤2.5×ULN, and in liver metastasis ≤5×ULN; serum bilirubin (TBIL) ≤1.5×ULN (except for Gilbert Syndrome ≤3×ULN); albumin (ALB) ≥30.0g/L (3) Renal function: serum creatinine ≤1.5×ULN or creatinine clearance rate (creatinine) ≤1.5×ULN. (3) Renal function: serum creatinine ≤1.5×ULN or creatinine clearance rate (CrCl) ≥50 mL/minute (using the Cockcroft/Gault formula) (4) Coagulation function: international normalized ratio (INR) ≤1.5; activated partial coagulation time (APCT) ≥1.5; activated partial coagulation time (APCT) ≤1.5 (4) Coagulation function: international normalized ratio (INR) ≤1.5, activated partial thromboplastin time (APTT) ≤1.5×ULN (5) Others: lipase ≤1.5×ULN; if lipase >1.5×ULN, the patient can be enrolled if there is no clinical or imaging evidence of pancreatitis; amylase ≤1.5×ULN; if amylase >1.5×ULN, the patient can be enrolled if there is no clinical or imaging evidence of pancreatitis; amylase ≤1.5×ULN; and amylase ≤1.5×ULN. or imaging evidence of pancreatitis can be enrolled. Alkaline phosphatase (ALP) ≤ 2.5 x ULN, and in subjects with bone metastases, ALP ≤ 5 x ULN (6) Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ 50%
10. Female patients who are non-surgically sterilized or of childbearing potential must have a negative serum HCG test within 72 hours prior to the first dose of study medication and must not be lactating, and must agree to use appropriate contraception (e.g., intrauterine device (IUD), birth control pills, or condoms) during the study treatment period and for 3 months after the end of the study treatment period; male patients must agree to use appropriate contraceptive methods during the study treatment period and for 3 months after the end of the study treatment period. Male patients agree to use an appropriate method of contraception during and for 3 months after study treatment.

Exclusion Criteria:

1. Patients with histologic or cytopathologic diagnosis of adenosquamous carcinoma or complex SCLC.
2. Genetic tests suggesting ALK fusion, ROS1 fusion, BRAF mutation, ERBB2 (HER2) amplification/mutation, RET rearrangement, MET amplification/MET14 exon jumping mutation and NTRK fusion positivity.
3. Clinical manifestations of neurologic failure such as severe encephalopathy or treatment-related severe neurologic injury, such as chemical meningitis
4. Non-malignant neurologic diseases that would interfere with the evaluation of LM signs or symptoms
5. radiotherapy directed to the chest and whole brain completed within 4 weeks prior to enrollment (palliative radiotherapy to bone lesions completed prior to the first dose of study drug is permitted for enrollment)
6. toxicity due to prior antitumor therapy other than alopecia and malaise not recovered to CTCAE 5.0 ≤ grade 1 prior to enrollment. Some other toxicities due to prior antitumor therapy are not expected to resolve within the expected period and have long-term persistent sequelae
7. patients with spinal cord compression that has not been cured or relieved by surgery and/or radiotherapy, or patients with previously diagnosed spinal cord compression that has been treated with compression insufficiency or total paralysis; patients with liver metastases who have received cryo- and radiofrequency ablation therapy and who still have clinically significant symptoms and abnormal hepatic function in the 4 weeks prior to enrollment
8. Presence of uncontrollable large amount of pleural effusion, pericardial effusion or ascites.
9. Presence of the following cardiac diseases: (1) cardiac function class III-IV according to NYHA cardiac function classification (2) unstable angina pectoris or electrocardiogram suggesting acute ischemia or myocardial infarction within 1 year (3) clinically significant supraventricular or ventricular arrhythmia and other conduction system abnormalities (including QTc interval greater than or equal to 450ms for men and ≥470ms for women) (4) clinically significant Pericardial and myocardial diseases
10. Inadequate bone marrow reserve or organ function
11. Treatment with systemic immunomodulators (including but not limited to thymidine, interferon, or interleukin-2) within 4 weeks prior to enrollment
12. Any active autoimmune disease or history of autoimmune disease; interstitial pneumonitis, drug-induced pneumonitis, radiation pneumonitis requiring steroid therapy, or active pneumonia with clinical symptoms
13. active or uncontrolled serious infection (CTCAE 5.0 ≥ grade 2) and/or antibiotic treatment within 2 weeks prior to enrollment
14. Patients with active or undergoing treatment for tuberculosis
15. Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg), history of hypertensive crisis or hypertensive encephalopathy
16. intracranial hemorrhage known to be unrelated to the tumor
17. imaging (CT or MRI) showing that the tumor invades large vessels or is poorly demarcated from them, or those who, in the opinion of the investigator, are predisposed to hemorrhage, with symptoms of hemoptysis or daily hemoptysis ≥ 2.5 mL within 3 months prior to screening
18. Have had an arterial/venous thrombotic event within 24 weeks prior to enrollment, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
19. Invasive surgery within 4 weeks prior to enrollment
20. Receiving medication with bleeding tendency, such as aspirin (>325 mg/day), or using full-dose oral or parenteral anticoagulants or thrombolytic agents for 2 weeks prior to enrollment.
21. Genetic predisposition to bleeding or coagulation disorders; clinically significant bleeding symptoms in the 12 weeks prior to enrollment or disorders with a clear bleeding predisposition, such as gastrointestinal bleeding, positive fecal occult blood at screening, or vasculitis.
22. History of peptic ulcer, gastrointestinal perforation, erosive esophagitis or gastritis, inflammatory bowel disease or diverticulitis, abdominal fistula, tracheo-esophageal fistula, or intra-abdominal abscess within 24 weeks prior to enrollment.
23. Urine routine suggests that urinary protein ≥++, and confirms that the quantitative amount of 24-hour urinary protein >1.0g
24. HBsAg positive and HBV DNA test value exceeds the upper limit of the normal reference value (1000 copies/mL or 100 IU/mL), or HCV positive (HCV RNA or HCV Ab test suggests acute and chronic infections); known history of HIV-positive disease.
25. Patients who have received a live vaccine within 12 weeks prior to enrollment
26. Known hypersensitivity to study drugs or excipients, known severe allergic reaction to any of the monoclonal antibodies
27. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
28. Other concurrent malignancies ≤ 5 years prior to the first dose of study drug, with the exception of adequately treatable carcinoma in situ of the cervix, basal cell or squamous epithelial skin cancers, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery
29. Known severe mental illness, alcoholism, drug addiction or drug abuse, etc.
30. Have been treated with any other experimental drug or participated in another interventional clinical study ≤ 4 weeks prior to signing the ICF.
31. In the judgment of the investigator, the subject has other factors that may lead to the forced termination of the study, such as non-compliance with the protocol, other serious illnesses (including psychiatric illnesses) that require co-treatment, serious laboratory abnormalities, associated family or social factors, which may affect the safety of the subject, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Two years of observation after enrollment
  Objective remission rates for flaccid meninges

SECONDARY OUTCOMES:
iPFS | Two years of observation after enrollment
  Intracranial progression-free survival
iDoR | Two years of observation after enrollment
  Duration of intracranial relief
PFS | Two years of observation after enrollment
  Overall progression-free survival
OS | Two years of observation after enrollment
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shengcun Fang, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No